CLINICAL TRIAL: NCT04365205
Title: Effect of Benralizumab on Airway Remodeling in Asthma
Acronym: BENRAMOD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/34
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Asthma
Keywords: Asthma; remodeling; IL-5 receptor; smooth muscle; biotherapy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchial specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- severe asthma: * Diagnosis of severe asthma according to the American Thoracic Society / European Respiratory Society task force.
  * Documented post-bronchodilator reversibility of at least 12% and at least 200 mL in Forced expiratory volume forced expiratory volume at one second (FEV1) within 12 months before enrollment.
  * Documented blood eosinophils ≥ 300 cells per μL within 12 months or blood eosinophils ≥150 cells per μL at visit 1.
  Interventions: Procedure: Endobronchial biopsy
- non-severe asthma: • Diagnosis of non-severe asthma according to the Global Initiative for Asthma (GINA).
  Interventions: Procedure: Endobronchial biopsy
- non-asthmatic controls: * No prior history of any chronic respiratory disease including asthma.
  * No prior history of allergy, i.e. allergic rhinitis, allergic conjunctivitis, hay fever, eczema.
  * No clinically significant abnormalities as determined by medical history, measurement of vital signs, physical examination, hematologic assessments and ECG at visit 1.
  * Normal lung function with FEV1 > 90%.
  Interventions: Procedure: Endobronchial biopsy

INTERVENTIONS:
Procedure: Endobronchial biopsy — Endobronchial biopsies will be collected following a standardized procedure based on established guidelines. Before the procedure, asthmatic subjects will receive 400 μg of salbutamol with the aid of an aerosol chamber to open up the airways before the procedure. Anesthesia of the upper airways will be achieved with lidocaine 5% spray. The total amount of lidocaine per subject is limited to 225 mg. General anesthesia will be obtained using propofol (average dose of 1.5 to 2 mg/kg). The fiberoptic bronchoscope (Pentax BF 15V, Argenteuil, France) is introduced and 8 to 10 biopsies will be taken from the middle lobe and the lower right lobe. Standard procedures such as bronchial brushing and bronchial fluid aspiration will also be performed. The duration of bronchoscopy is 15 minutes to 30 minutes. After the procedures, subjects will receive a short acting bronchodilator if required.

SUMMARY:
The anti-interleukin (IL)-5 receptor benralizumab inhibits eosinophilic inflammation but its potential effect on airway remodeling remains unknown. The main objective of this study is to assess the effect of benralizumab in an in vitro model of airway remodeling using cells obtained from asthmatic patients.

DETAILED DESCRIPTION:
Sixty subjects will be recruited: 20 patients with severe asthma patients, 20 patients with non-severe asthma and 20 non-asthmatic controls. Inclusion visit will include written informed consent, asthma questionnaire, clinical examination, lung function testing, prick tests and assessment of airway remodeling using CT scan and MRI. Bronchial specimens from all subjects will be obtained by fiberoptic bronchoscopy. Airway remodeling will be evaluated by morphological analysis. After BSM cell culture, BSM cells function will be assessed in vitro in the absence or presence of benralizumab using proliferation (BrdU) and chemotactism experiments, ELISA, RT-PCR (polymerase chain reaction ) and electronic microscopy.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* Written informed consent indicating that they understand the purpose and procedures required for the study and are willing to participate in the study.
* Age higher than 18 years.
* No prior history of any chronic respiratory disease including asthma.
* No prior history of allergy, i.e. allergic rhinitis, allergic conjunctivitis, hay fever, eczema.
* No clinically significant abnormalities as determined by medical history, measurement of vital signs, physical examination, hematologic assessments and ECG at visit 1.
* Normal lung function with FEV1 > 90%.

Non-severe asthmatics subjects

* • Written informed consent indicating that they understand the purpose and procedures required for the study and are willing to participate in the study.
* Age higher than 18 years.
* Diagnosis of non-severe asthma according to the Global Initiative for Asthma (GINA), i.e. GINA steps 1, 2 or 3 (18).
* Documented post-bronchodilator reversibility of at least 12% and at least 200 mL in FEV1 within 12 months before enrolment, or PC20 methacholine < 16 mg/mL documented within 12 months prior to screening.
* Documented blood eosinophils ≥300 cells per μL within 12 months or blood eosinophils ≥150 cells per μL at visit 1.

Severe asthmatics subjects

* • Written inform consent indicating that they understand the purpose and procedures required for the study and are willing to participate in the study.
* Age higher than 18 years.
* Diagnosis of severe asthma according to the American Thoracic Society (ATS)/European Respiratory Society (ERS) task force (19).
* Documented post-bronchodilator reversibility of at least 12% and at least 200 mL in FEV1 within 12 months before enrolment.
* Documented blood eosinophils ≥300 cells per μL within 12 months or blood eosinophils ≥150 cells per μL at visit 1.

Exclusion Criteria:

* Active smoker or former smoker.
* Diagnosis of chronic obstructive pulmonary disease (COPD), cystic fibrosis, or other significant respiratory disorder including significant occupational or environmental exposures with ongoing respiratory symptoms.
* CT scan abnormality related to any respiratory disease other than asthma.
* Recent asthma exacerbation (less than 6 weeks before bronchoscopy).
* Contraindications related to bronchoscopy:

  * coagulation disorders,
  * unstable cardiovascular conditions,
  * FEV1 lower than 1 litter,
  * a fasting state of less than 6 hours for food and less than 2 hours for drink.
* Contraindications to general anesthesia or medications (for propofol: hypersensitivity to the active substance and to any of the excipients; for lidocaine: hypersensitivity to the active substance and to any of the excipients or to local anesthetics of the amide type, epilepsy, porphyria) used in the bronchoscopy procedure.
* Contraindications related to MRI:

  * Pacemaker or implantable cardioverter defibrillator
  * Metallic foreign body in the eye
  * Cerebral aneurysm clips
  * Insulin pumps
  * Claustrophobia
* Positive urinary pregnancy test at screening for women of child-bearing potential
* Breastfeeding woman.
* Previously received benralizumab.
* History of any clinically significant medical illness or medical disorders including (but not limited to) cardiovascular disease, neuromuscular, hematological disease including bleeding disorders, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease.
* Recent history (within previous 6 months) of alcohol or drug abuse.
* Persons placed under judicial protection.
* Persons participating in another research including a period of exclusion still in course.
* Severely altered physical and/or psychological health which, according to, the investigator, could affect the participant's compliance of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects with no prior history of any chronic respiratory disease including asthma (n = 20), non-severe asthmatics subjects (n = 20) and severe asthmatics (n = 20).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-10-05 (Estimated); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
Number of Bronchial smooth muscle (BSM) cells obtained from severe asthmatics measured in vitro using BrdU incorporation. | Month 12
  Determine the proliferation of BSM cells obtained from severe asthmatics measured in vitro using BrdU incorporation.

SECONDARY OUTCOMES:
Number of cultured BSM cell from non-severe asthmatics and healthy volunteers measured using BrdU incorporation. | Month 12
  Determine the proliferation of cultured BSM cell from non-severe asthmatics and healthy volunteers measured using BrdU incorporation.
Number of different genes | Month 12
  Gene expression within BSM cells (RT-PCR, nCCounter Immunology panels)
Measure the inflammatory mediators and extracellular components | Month 12
  Production of inflammatory mediators and extracellular components by cultures BSM cells (ELISA, bio-Plex® Multiples Immunoassays)
Measure the fluorescence intensity of IL-5 receptor subunit alpha on BSM cells | Month 12
  Determine of expression of IL-5 receptor subunit alpha on BSM cells (% of positive cells, mean fluorescence intensity) using flow cytometry
Count the number of mitochondria / BSM area (x107/mm2) | Month 12
  Determine of number of mitochondria / BSM area (x107/mm2) and mitochondrial density using electron microscopy
Count the number of eosinophils/smooth muscle area using optic microscopy | Month 12
  Histological criteria: BSM area (% of tissue area), number of eosinophils/smooth muscle area using optic microscopy
Measure the bronchial dimension by CT-scan | Month 12
  Bronchial dimensions assessed by CT-scan
Measure the bronchial dimension by MRI | Month 12
  Bronchial dimensions assessed by MRI
Measure the lung low single intensity and low attenuation values using MRI | Month 12
  Determine the Lung low single intensity and low attenuation values using MRI
Measure the lung low single intensity and low attenuation values using CT-scan | Month 12
  Determine the Lung low single intensity and low attenuation values using CT-scan

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Olivier GIRODET, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CIC-P - Centre François Magendie - G3 - Hôpital Haut-Lévêque, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No